CLINICAL TRIAL: NCT01551693
Title: This Trial is an Open Label, Parallel Cohort, Phase II Study Evaluating the Efficacy of the Heat Shock Protein 90 (Hsp90) Inhibitor STA-9090 in Patients With Unresectable Stage III or Stage IV Melanoma Who Were Intolerant of, or Progressed on, Prior Tyrosine Kinase Inhibitor Treatment. Two Cohorts Will Enroll Concurrently. One Cohort Will be Composed of Patients With Melanoma Expressing a Mutation in the Protein BRAF and the Other Cohort Will be Composed of Patients With Melanoma Expressing Wild-type BRAF.
Brief Title: STA-9090(Ganetespib) in Patients With Unresectable Stage III or Stage IV Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: due to weak accrual
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Synta Pharmaceuticals Corp. (Industry)
Responsible Party: Principal Investigator, F. Stephen Hodi, MD, Melanoma Disease Center Director, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-039
Record Dates: First submitted 2011-04-29; First posted 2012-03-13 (Estimated); Results first posted 2017-04-12 (Actual); Last update posted 2017-04-12 (Actual); Status verified 2017-01

CONDITIONS: Melanoma
Keywords: Stage III; Stage IV; Unresectable; Metastatic
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis | interventions — STA 9090

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- STA-9090 Cohort A (Experimental): Patients enrolled into two possible cohorts based on tumor expression of BRAF: Cohort A - BRAF mutant disease or Cohort B - BRAF wild type. Cohort A patients received STA-9090 200 mg/m2 once weekly (d1, 8, 15 of 28 day cycle). Patients were treated until evidence of disease progression, unacceptable toxicity, intercurrent illness or withdrawal.
  Interventions: Drug: STA-9090
- STA-9090 Cohort B (Experimental): Patients enrolled into two possible cohorts based on tumor expression of BRAF: Cohort A - BRAF mutant disease or Cohort B - BRAF wild type. Cohort B patients received STA-9090 150 mg/m2 twice weekly (d1, 4, 8, 11, 15, 18 of 28 day cycle). Patients were treated until evidence of disease progression, unacceptable toxicity, intercurrent illness or withdrawal.
  Interventions: Drug: STA-9090

INTERVENTIONS:
Drug: STA-9090
  Other Names: Ganetespib

SUMMARY:
STA9090 is a drug which inactivates or blocks the work of a protein called Heat Shock Protein 90 or HSP90. HSP90 is a protein that helps some molecules inside your cells to have the right shape. By stopping HSP90's activity, those molecules never get to have the right structure of be functional and they are destroyed. The investigators believe that if they stop the activity of HSP90, the rapidly dividing cells that are in your tumor(s) may slow down. In this research study the investigators are looking to see how well STA9090 works in stopping the spread of your melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the proportion of patients alive, free of disease progression, and still taking STA-9090 at 6 months by BRAF mutant or wild type (WT) status.

Secondary

* To assess best overall response rate and six month response rate by BRAF status
* To evaluate the rates of one-year overall survival and progression-free survival by BRAF status
* To determine safety and tolerability of STA-9090 by BRAF status

Exploratory

* To compare the rates of response and of six-month PFS between BRAF status cohorts
* To explore, using peripheral blood mononuclear cells, the relationship between change in expression of hsp90 client proteins (e.g., BRAF, CRAF, AKT, CDK4, KIT) with response to therapy and progression free survival by BRAF status
* To explore the relationship in biopsied melanoma metastases between changes in expression of hsp90 client proteins (e.g., BRAF, CRAF, AKT, CDK4, KIT) with response to therapy and progression-free survival
* To explore response rate and 6 month progression free survival, in subset of patients with melanoma expressing a mutation in KIT

ELIGIBILITY:
* Histologically confirmed unresectable stage III or stage IV melanoma
* Treatment of unresectable stage III or stage IV melanoma with a tyrosine kinase inhibitor within prior 4 months. Sorafenib for purposes of eligibility will not be considered acceptable prior therapy
* Sufficient tumor available to determine if expresses wild-type or mutated BRAF if result not already known. The presence or absence of BRAF mutation needs to be determined at BWH, MGH, BIDMC, by Drs. Christopher Corless and Michael Heinrich at Cancer Pathology Shared Resource Oregon Health & Science University, or in context of eligibility assessment after signing consent to a previous clinical trial
* Sufficient tumor available to determine if expresses a mutation KIT
* Agreement to allow tumor to be evaluated for mutations in KIT and BRAF
* ECOG performance status ≤ 1
* Life expectancy of ≥ 6 months
* Age ≥ 18 years
* WBC ≥ 3 x 103/ul
* ANC ≥ 1,500/ul
* Platelets ≥ 100 x 103/ul
* Hemoglobin ≥ 9 gm/dl
* Serum creatinine ≤ 1.5 x ULN
* Calculated creatinine clearance ≥ 60 mL/min
* AST ≤ 2.5 x ULN; -OR- AST ≤ 5 x ULN in the presence of known liver metastases
* ALT ≤ 2.5 x ULN; -OR- ALT ≤ 5 x ULN in the presence of known liver metastases
* Total bilirubin ≤ 1.5 x ULN
* Potassium within normal range or correctable with supplements
* Magnesium within normal range or correctable with supplements
* Corrected serum calcium within normal range, or correctable with supplements
* Not pregnant or breastfeeding. Female subjects of childbearing age must have a negative serumpregnancy test at study entry
* Women of childbearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation and for 6 months following last study drug administration
* Agreement to provide blood samples for pharmacodynamic studies utilizing Peripheral Blood Mononuclear Cells (PMBCs) as outlined in protocol
* At least one site of measurable disease as defined by at least 1 cm in greatest dimension. This site must be different from the sites to be used for biopsy. No prior radiation therapy or directed ablation to the site of measureable disease
* Able to understand and willing to sign a written informed consent document
* Willing and able to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures
* No chemotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to study entry
* No radiotherapy within 4 weeks prior to study entry
* Subject has recovered from adverse events due to agents administered more than 4 weeks earlier
* No tyrosine kinase inhibitor within 14 days prior to study entry
* No major surgery within 4 weeks prior to first dose of STA-9090
* No minor surgery within 7 days of first dose of STA-9090
* No history of or current coronary artery disease, myocardial infarction, angina pectoris, angioplasty
* or coronary bypass surgery
* No current treatment with the following antiarrythmic drugs: flecainide, moricizine or propafenone
* No NYHA class II/III/IV congestive heart failure with a history of dyspnea, orthopnea, or edema that requires current treatment with angiotensin convering enzyme inhibitors, angiotensin II receptor blockers, beta-blockers, or diuretics
* No current or prior radiation to the left hemithorax
* No embolization procedure or ablation procedure to treat tumor within 4 weeks of first dose of STA- 9090
* Not receiving any other investigational agents
* No poor venous access for study drug administration unless subject can use silicone based catheters
* No history of brain metastases or of leptomeningeal involvement
* No history of severe allergic reactions or hypersensitivity reactions attributed to compounds of similar chemical or biologic composition to STA-9090 (e.g. olyethylene glycol [PEG] 300 or Polysorbate 80)
* Baseline QTc ≤ 470 msec
* No previous history of QT prolongation while taking other medications
* Ventricular ejection fraction (EF) > 55%
* No treatment with chronic immunosuppressants
* No melanoma of ocular primary
* No prior treatment with hsp90 inhibitor
* No uncontrolled intercurrent illness including, but not limited to ongoing or active infection, ventricular arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* No other medications, or severe acute/chronic medical of psychiatric conditions or laboratory abnormality that may increase the risk associated with the study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the subject inappropriate for entry into the study
* No history of a different malignancy except for the following circumstances. Individuals with a history of other malignancies are eligible if they have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin
* No HIV-positive subject on combination antiretroviral therapy
* No more than 3 prior systemic therapies for unresectable stage III or stage IV melanoma
* No concomitant use of medications associated with a high incidence of QT prolongation as outlined

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: F. Stephen Hodi, M.D., Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients enrolled from September 2011 to March 2012.
Period: Overall Study
Arm/Group | STA-9090 Cohort A | STA-9090 Cohort B
Started | 1 | 2
Completed | 0 | 0
Not Completed | 1 | 2
Not completed — Disease Progression | 1 | 0
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: The analysis dataset is comprised of all treated patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | STA-9090 Cohort A | STA-9090 Cohort B | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Continuous [Mean (Full Range); unit: years] | 60 [60 to 60] | 75 [68 to 83] | 71 [60 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: 6-month Progression-Free Survival Rate
Description: 6-month progression-free survival rate was defined as the proportion of patients absent death or progression based on Response Evaluation Criteria In Solid Tumors Criteria (RECIST) before 6 months. Per RECIST 1.0 criteria: progressive disease (PD) is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. PD for the evaluation of non-target lesions is the appearance of one or more new lesions and/or unequivocal progression of non-target lesions.
Time Frame: Disease was evaluated radiologically at baseline and every 8 weeks on treatment; Treatment continued until evidence of disease progression or unacceptable toxicity. Relevant for this endpoint was disease status at 6 months.
Measure: Number; unit: proportion of participants
Arm/Group | STA-9090 Cohort A | STA-9090 Cohort B
Number analyzed (Participants) | 1 | 2
proportion of participants | 0.0 | 0.0

2. Secondary Outcome: Best Overall Response
Description: Best overall response (BOR) on treatment was based on RECIST 1.0 criteria. For target lesions, complete response (CR) is complete disappearance of all target lesions and partial response (PR) is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. CR or PR confirmation required within 4 weeks. Progressive disease (PD) is at least a 20% increase in the sum LD of target lesions from smallest sum LD as reference or the appearance of one or more new lesions. Stable disease (SD) is neither meeting PR or PD. PD for the evaluation of non-target lesions is the appearance of one or more new lesions and/or unequivocal progression of non-target lesions. CR is disappearance of all non-target lesions.
Time Frame: Disease was evaluated radiologically at baseline and every 8 weeks on treatment. Median (range) treatment duration was 1 cycle/4 weeks (1-2 cycles; 4-8 weeks).
Measure: Number; unit: participants
Arm/Group | STA-9090 Cohort A | STA-9090 Cohort B
Number analyzed (Participants) | 1 | 2
participants
  Progressive Disease | 1 | 1
  Unevaluable | 0 | 1

3. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from study entry to death or date last known alive and estimated using Kaplan-Meier (KM) methods.
Time Frame: Patients were followed every 4 weeks for survival until death, lost to follow-up or study closure (approximately 6 months after the last patient ended treatment). In this study cohort, patients were followed up to 13 weeks.
Population: Overall survival was not estimated given the limited sample size.
Arm/Group | STA-9090 Cohort A | STA-9090 Cohort B
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: AE assessment was ongoing from the start of study drug and up to day 30 post-treatment. Mean treatment duration was 1 cycle/4 weeks (range 1-2 cycles/4-8 weeks).
Description: Maximum grade toxicity by type was first calculated. Serious AEs were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher per CTCAEv3. Other AEs were defined as events with treatment-attribution of possible, probable or definite and grades 1 or 2 per CTCAEv3.
Arm/Group | STA-9090 Cohort A | STA-9090 Cohort B
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/2
Other Adverse Events (participants affected / at risk) | 0/1 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | STA-9090 Cohort A (N=1) | STA-9090 Cohort B (N=2)
Alkaline phosphatase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | STA-9090 Cohort A (N=1) | STA-9090 Cohort B (N=2)
Anemia (Blood and lymphatic system disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The study was terminated early due to weak accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No